CLINICAL TRIAL: NCT03114293
Title: Evidence Based Patient Information and Smartphone Accelerometry to Enhance Physical Activity in MS
Acronym: PIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Jan-Patrick Stellmann, MD, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: inims-pia
Record Dates: First submitted 2017-03-31; First posted 2017-04-14 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis, Chronic Progressive
Keywords: Physical activity; Mobility
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Motor Activity

STUDY DESIGN:
Intervention Model Description: Short, randomised waiting-group controlled explorative studies of a behavioural intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Rater blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waiting group (No Intervention): Waiting group
- Smartphone intervention (Experimental): Smartphone bases behavioural intervention
  Interventions: Behavioral: Smartphone App

INTERVENTIONS:
Behavioral: Smartphone App — The app includes an EBPI and physical activity feedback
  Arms: Smartphone intervention

SUMMARY:
Due to their ubiquitary distribution, smartphones might serve as an easy way/ possibility to use feedback mechanism in an app-based intervention program to increase physical activity in Multiple Sclerosis (MS) patients. Internet based cognitive-behavioral interventions have been explored as effective in the last years. In addition, smartphone-based mobility assessment and intervention might be a promising approach in other MS types and for real-life mobility assessment in observational and interventional trials. The aim is to investigate the impact of a smartphone based information and feedback program on physical activity in a 3 months, randomised waiting-group controlled trial of 40 progressive MS patients.

ELIGIBILITY:
Inclusion Criteria:

* progressive MS

Exclusion Criteria:

* other major health disorder
* EDSS above 6

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-05-30 (Estimated); Study Completion 2017-05-30 (Estimated)

PRIMARY OUTCOMES:
Rate of responders | 3 Months
  Rate of responders as defined by a 20% increase of steps or 20% increase in physical activity as measured with the actigraph

SECONDARY OUTCOMES:
Physical activity: total activity | 3 Months
  Physical activity and real-life mobility: 1-week accelerometry (actigraph)
Physical activity: distance per day | 3 Months
  Physical activity and real-life mobility: 1-week accelerometry (actigraph)
Physical activity: number of steps per day | 3 Months
  Physical activity and real-life mobility: 1-week accelerometry (actigraph)
Questionnaires on quality of life (QoL, HAQUAMS) | 3 Months
  Disease specific quality of life questionnaire
Questionnaires on activities of daily living (ADL) | 3 Months
  Frenchay activity index
Questionnaires on physical activity | 3 Months
  Godin Leisure time

IPD SHARING:
Plan to Share IPD: Undecided